CLINICAL TRIAL: NCT05046184
Title: Elucidating the Neurocircuitry of Irritability With High-Field Neuroimaging to Identify Novel
Brief Title: Elucidating the Neurocircuitry of Irritability With High-Field Neuroimaging to Identify Novel Therapeutic Targets
Acronym: UNIKET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Manish Jha, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: STU-2021-0667
Record Dates: First submitted 2021-08-23; First posted 2021-09-16 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder; Healthy Controls
Keywords: major depressive disorder; MDD; depression; depressive disorder; depression symptoms; healthy controls; irritability; ketamine
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder | interventions — Ketamine; Midazolam

STUDY DESIGN:
Intervention Model Description: All subjects (Healthy Controls and MDD) will undergo resting-state and task-based fMRI and cerebral prefusion to characterize the (i) patterns of functional connectivity and (ii) neural responses to a behavioral task eliciting frustrative nonreward (FNR) that are associated with irritability [quantified with the 5-item irritability domain of Concise Associated Symptom Tracking scale (CAST-IRR)]. The MDD cohort (n=60) will then be randomized to four 40-minute intravenous infusions over two weeks of either ketamine (0.5 mg/kg) or midazolam (0.02 mg/kg) in a double-blind, parallel-arm fashion. Clinical assessments and 3T MRI scans will be repeated after the last infusion to evaluate (i) pre-to-post treatment changes in neurocircuit function using resting-state and FNR task-based fMRI with ketamine versus midazolam and (ii) the association between changes in neurocircuit function and irritability.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects and study team members, including the PI, study-affiliated physicians, coordinator, nursing staff, and data analysts will be blinded to the drug assignment until the completion of the proposed project. Only the research pharmacist and study members involved in safety monitoring (medical monitor, independent safety monitor, and data analyst responsible for generating safety reports) will know the identity of the drug.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Healthy Controls (No Intervention): Healthy controls will undergo clinician assessments and fMRI to compare to MDD group.
- MDD - Ketamine (Active Comparator): Participants with MDD who have completed all baseline assessments including pre-treatment fMRI scan randomly allocated to receive four ketamine infusions.
  Interventions: Drug: Ketamine Hydrochloride
- MDD - Midazolam (Placebo Comparator): Participants with MDD who have completed all baseline assessments including pre-treatment fMRI scan randomly allocated to receive four midazolam infusions.
  Interventions: Drug: Midazolam injection

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Subjects with MDD will receive 2 weeks of twice-weekly 40-minutes long IV infusion of ketamine (0.5 mg/kg). Ketamine will be dissolved in 0.9% saline in a total volume of 100 mL and administered with an infusion pump at a constant rate.
  Arms: MDD - Ketamine
Drug: Midazolam injection — Subjects with MDD will receive 2 weeks of twice-weekly 40-minutes long IV infusion of midazolam (0.02 mg/kg). Midazolam will be dissolved in 0.9% saline in a total volume of 100 mL and administered with an infusion pump at a constant rate.
  Arms: MDD - Midazolam

SUMMARY:
The study is investigating dysfunctions in neurocircuitry in regards to irritability with healthy controls (HC) and individuals with Major Depressive Disorder (MDD) by performing MRIs. The MDD group will also be randomized to receive ketamine or midazolam to investigate changes post-treatment in neurocircuitry with regards to irritability.

DETAILED DESCRIPTION:
The proposed study aims to 1 (Aim 1) identify dysfunctions in neurocircuitry that engender irritability, and (Aim 2) determine how changes in neurocircuit function related to change in irritability. We will accomplish Aim 1 with resting-state and frustrative nonreward (FNR) task-based fMRI data from n=30 HCs and n=60 subjects with MDD ((Fig 3). For Aim 2, we will randomize the MDD cohort (n=60; same as Aim 1) to 2 weeks of twice-weekly 40-minutes long intravenous infusion of either ketamine (0.5 mg/kg) or midazolam (0.02 mg/kg) in a double-blind parallel-arm fashion, and by repeating clinical assessments and fMRI scans after the last infusion. The central hypothesis of the proposed study is that striatum is a key hub in the neurocircuitry of irritability, and that treatment-related improvement in irritability is associated with normalization of these neurocircuit functioning.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 18-65 years of age and body weight less than or equal to 120 kg on baseline visit.
2. Participants must have a level of understanding of the English language sufficient to agree to all tests and examinations required by the study and must be able to participate fully in the informed consent process.
3. For Healthy Controls: Subjects must be free of any lifetime psychiatric condition based on the Mini-International Neuropsychiatric Interview (MINI). For MDD: Subjects must meet Diagnostic and Statistical Manual of Mental Disorders (DSM-5) criteria for current unipolar depression [major depressive disorder (MDD) or persistent depressive disorder (PDD) in a current major depressive episode (MDE)] based on MINI.
4. A woman of childbearing potential who is sexually active with a male must agree to use an acceptable method of contraception [defined as either one highly effective (permanent sterilization, intrauterine device or hormonal implant) or two other forms of contraception (such as oral contraceptive pill and condom)] to avoid pregnancy throughout the study. Throughout the study and for 90 days (one spermatogenesis cycle) after receiving the last dose of study drug (ketamine/midazolam) man who is sexually active with a woman of childbearing potential must use an acceptable method of contraception (described above) with his female partner and must agree not to donate sperm.
5. Subjects must either be free of psychotropic medications (including antidepressants, antipsychotics, benzodiazepines, mood stabilizers, sedative/hypnotics, dopamine agonists, stimulants, buspirone, and triptans) and certain anticonvulsants (topiramate and levetiracetam) or be stable on these medications for four weeks prior to the baseline visit [first magnetic resonance imaging (MRI) scan].
6. Subjects with MDD should be willing to participate in neuroimaging scans before and after infusions, and be willing to undergo infusions with study drug.

Exclusion Criteria:

1. Lifetime diagnosis of schizophrenia or any psychotic disorder, bipolar disorder, pervasive developmental disorder or intellectual development disorder.
2. Current diagnosis of obsessive-compulsive disorder, anorexia nervosa or bulimia. Comorbid anxiety, stress and trauma-related disorders are permitted as long as unipolar depression is the primary diagnosis.
3. Diagnosis of a moderate or severe substance use disorder within the past 6 months per MINI; all subjects must have a negative urine toxicology test on the day of the MRI, prior to the scan.
4. Female subjects who are pregnant, nursing, for may become pregnant. Women of childbearing potential must have a negative urine pregnancy test on the day of the fMRI, prior to scan, and on days of study drug infusion, prior to infusion.
5. Any unstable medical illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, immunologic, or hematologic disease.
6. Inadequately treated obstructive sleep apnea (STOP-Bang score of 5-8 if untreated, if using positive airway pressure device then past-month apnea hypopnea index ≥ 15 per hour representing moderate or higher severity).
7. Presence of a significant neurological disease such as Parkinson's disease, primary or secondary seizure disorders, intracranial tumors, or severe head trauma.
8. Presence of neurocognitive or dementing disorders.
9. Clinically significant abnormalities of laboratories, physical examination (including unstable hypertension - systolic blood pressure >170, diastolic blood pressure >100), or electrocardiogram at screening visit.
10. Subjects judged to be at serious and imminent suicidal or homicidal risk by the PI or another study-affiliated psychiatrist.
11. Any contraindications to MRI, including pacemakers or metallic objects in the body.
12. Any claustrophobia or other conditions which may result in inability to lie still in the MRI scanner for 1 hour or more.
13. Allergy to ketamine or midazolam in subjects with MDD.
14. Must not be on any prohibited concomitant medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Resting state functional connectivity. | Baseline
  Resting-state functional connectivity between striatum and habenula will be measured by functional magnetic resonance imaging (fMRI) in healthy controls and in adults with major depressive disorder (MDD). Functional connectivity refers to the standardized correlation between resting state BOLD signal of the striatum and habenula regions of the brain.
Striatal response to frustrative nonreward (FNR). | Baseline
  Striatal response to frustrative nonreward (FNR) as measured by the BOLD (Blood Oxygen Level Dependent) signal within the striatum region of the brain on a functional MRI behavioral task of FNR in healthy controls and in adults with MDD. BOLD signal is the unit of measure of this outcome.
Treatment-related change in striatum-habenula functional connectivity. | Baseline, at 14 days
  Striatum-habenula functional connectivity is the standardized correlation between resting state BOLD signal of the striatum and habenula regions of the brain measured on a fMRI. Unit is the standardized correlation ranges from -1 to 1. MDD participants only.
Treatment-related change in striatal response to FNR. | Baseline, at 14 days
  Striatal response to FNR is the standardized correlation between resting state BOLD signal of the striatum and habenula regions of the brain measured on a fMRI. Unit is the standardized correlation ranges from -1 to 1. MDD participants only.

SECONDARY OUTCOMES:
Change in symptoms of irritability after two weeks of twice-weekly infusions of ketamine versus midazolam. | Baseline, at 14 days
  Symptoms of irritability will be measured by Concise Associated Symptom Tracking scale (CAST-IRR) where possible scores range from 5-25 and higher scores indicate greater severity of irritability. MDD participants only.
Change in symptoms of depression (including suicidal ideation) measured by MADR scale | Baseline, at 14 days
  Symptoms of depression will be measured by Montgomery-Åsberg Depression Rating Scale (MADRS). Possible scores range from 0 to 60 where higher scores indicate worse outcome. MDD participants only.
Change in symptoms of depression measured by QIDS report | Baseline, at 14 days
  Symptoms of depression will be measured by Quick Inventory of Depressive Symptomatology (QIDS) report. Possible scores range from 0 to 27 where higher scores indicate worse outcome. MDD participants only.
Change in symptoms including anxious arousal measured by MAS questionnaire | Baseline, at 14 days
  Symptoms including anxious arousal will be measured by Mood and Anxiety Symptoms Questionnaire (MASQ). Possible scores range from 1-5 where higher scores indicate worse outcome. MDD participants only.
Change in behavior (including anger attacks) measured by AAQ | Baseline, at 14 days
  Behavior (including anger attacks) will be measured by Massachusetts General Hospital Anger Attack Questionnaire (AAQ) as 'Yes/No' where 'Yes' means worse outcome. MDD participants only. MDD participants only.
Change in severity of dissociative symptoms associated with study drug administration measured by CADS scale | Baseline, at 14 days
  Severity of dissociative symptoms associated with study drug administration (Ketamine vs Midazolam) will be measured by Clinician-Administered Dissociative States Scale (CADSS). Possible scores range from 0-5 where higher scores indicate worse outcome. MDD participants only
Change in patient reported side effects measured by PRISE Adverse Event scores | Baseline, at 14 days
  Patient reported side effects will be measured by Patient Rated Inventory of Side Effects (PRISE) Adverse Event visit checklist. The PRISE is a physician-administered checklist of adverse events. PRISE contains 33 items, each defined by an adverse event. Each item is rated on a 3-point scale, ranging from 0 (not present) to 2 (distressing), with a total score range from 0-66, where higher scores indicate more adverse events. MDD participants only
Acute behavioral changes measured by Brief Psychiatric Rating Scale (BPRS) | Baseline, at 14 days
  Acute behavioral changes will be measured by Brief Psychiatric Rating Scale (BPRS) that consists of 18 items, each defined by a series of symptoms. Each item is rated on a 7-point scale, ranging from 1 (not observed) to 7 (very severe), with a total score range from 18-126, where higher scores indicate psychiatric symptoms. MDD participants only

OTHER OUTCOMES:
To evaluate if changes in neurocircuit function with ketamine mediate treatment-related improvement in irritability. | Up to 14 days
  Exploratory analyses will also evaluate neurocircuit mechanisms using measures of cerebral perfusion.

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States